CLINICAL TRIAL: NCT04647461
Title: Comparison of Efficacy and Ocular Surface Disease Assessment Between BRIDIN-T Eye Drops 0.15% and ALPHAGAN-P Eye Drops 0.15% in Glaucoma or Ocular Hypertensive Patients : Phase 4, Parallel Group Design, Investigator-blind, Active-control, Randomized, Multi-center Trial
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: CHA University (Other)
Collaborators: Hanlim Pharm. Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Seungsoo Rho, Associate Professor., M.D., Ph.D., CHA University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BAT
Record Dates: First submitted 2020-11-23; First posted 2020-12-01 (Actual); Last update posted 2020-12-01 (Actual); Status verified 2020-11

CONDITIONS: Glaucoma; Ocular Hypertensive
MeSH Terms: conditions — Glaucoma | interventions — Brimonidine Tartrate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BRIDIN-T Eye drops 0.15%(Non preservative) (Experimental): Brimonidine Tartrate 1.5mg : 1 drop 3 times a day for 12 weeks to target eyes
  Interventions: Drug: Brimonidine Tartrate 1.5mg
- ALPHAGAN-P Eye drops 0.15%(Preservatives) (Active Comparator): Brimonidine Tartrate 1.5mg : 1 drop 3 times a day for 12 weeks to target eyes
  Interventions: Drug: Brimonidine Tartrate 1.5mg

INTERVENTIONS:
Drug: Brimonidine Tartrate 1.5mg — 1 drop 3 times a day for 12 weeks to target eyes
  Other Names: BRIDIN-T Eye drops 0.15%
  Arms: BRIDIN-T Eye drops 0.15%(Non preservative)
Drug: Brimonidine Tartrate 1.5mg — 1 drop 3 times a day for 12 weeks to target eyes
  Other Names: ALPHAGAN-P Eye drops 0.15%
  Arms: ALPHAGAN-P Eye drops 0.15%(Preservatives)

SUMMARY:
Comparison of Efficacy and Ocular Surface Disease Assessment between BRIDIN-T Eye drops 0.15% and ALPHAGAN-P Eye drops 0.15% in Glaucoma or Ocular Hypertensive Patients : Phase 4, Parallel Group Design, Investigator-blind, Active-control, Randomized, Multi-center Trial

DETAILED DESCRIPTION:
Following 12 weeks of administration of BRIDIN-T Eye drops 0.15%(non preservative) or ALPHAGAN-P Eye drops 0.15%(preservatives) for patients with glaucoma or Ocular Hypertensive Patients. The use of BRIDIN-T Eye drops(non preservative) is less harmful to external ophthalmicus diseases and increase of medication compliance for ophthalmic drugs than the ALPHAGAN-P Eye drops 0.15%(preservatives)

ELIGIBILITY:
Inclusion Criteria:

1. Adult(Male or Female) over 19 years who were diagnosed with glaucoma or ocular hypertension
2. In the case of a person receiving a glaucoma treatment drug, a person who has completed the appropriate in wash-out period for the existing glaucoma drug before the investigational product is administered.
3. Intraocular pressure (IOP) >/= 15mmHg and < 40mmHg in each eye using Goldmann applanation tonometry at visit 2
4. Written consent voluntarily to participate in this clinical trial

Exclusion Criteria:

1. Patients with primary closed-angle glaucoma, congenital glaucoma and secondary glaucoma caused by steroid drugs, etc.
2. BCVA (best-corrected visual acuity) Snellen equivalent of Snellen 20/80(logMar 0.25) or less.
3. Those who have ongoing medical history as intraocular inflamation.
4. Central corneal thickness is not between 470um and 591um.
5. Patients who have received lacrimal passive occlusion within the last three months or who have surgery plans during the clinical trial period.
6. Pregnant or nursing women.
7. Patients judged coexisting disease that could interfere with the completion of the treatment or safety of this clinical trial. Patients that other researchers are determined inadequately

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2019-03-20 (Actual); Primary Completion 2021-01-29 (Estimated); Study Completion 2021-01-29 (Estimated)

PRIMARY OUTCOMES:
Corneal staining test | Administered 12 weeks after
  The degree of staining of the cornea after blue fluorescein staining under the slit lamp illumination of a cobalt blue light source using a yellow filter was evaluated on a 6 point scale according to the oxford grading system
Conjunctival staining test | Administered 12 weeks after
  After lysamine green staining under slit lamps, the conjunctiva was divided into the nasal side and the lateral side, and the degree of nasal conjunctiva and bilateral conjunctival staining was evaluated on a 6-point scale according to the oxford grading system
Ocular surface disease index (OSDI) | Administered 12 weeks after
  The ocular surface disease index was assessed for ocular surface disease, including visual function (five items), eye symptoms (four items), and environmental factors (three items) , 0 point for no symptoms, 1 point for occasional symptoms, 2 points for symptoms of half a day, 3 points for most symptoms, and 4 points for symptoms during the whole day.
Questionnaire (Evaluation of Satisfaction with Medication, Ocular tolerance) | Administered 12 weeks after
  The evaluation of satisfaction with medication is conducted with a questionnaire evaluation on the convenience of use, storage of investigational product, and the ocular tolerance.
  Evaluation is conducted on 8 symptoms of tingling/hot, sticky, itchy, blurred vision, foreign body sensation, dryness, glare, and pain. Assess the severity of symptoms (0-3 points) and duration of symptoms (immediate, continuous)

SECONDARY OUTCOMES:
Corneal staining test | Administered 4 weeks after
  The degree of staining of the cornea after blue fluorescein staining under the slit lamp illumination of a cobalt blue light source using a yellow filter was evaluated on a 6 point scale according to the oxford grading system
Conjunctival staining test | Administered 4 weeks after
  After lysamine green staining under slit lamps, the conjunctiva was divided into the nasal side and the lateral side, and the degree of nasal conjunctiva and bilateral conjunctival staining was evaluated on a 6-point scale according to the oxford grading system
Ocular surface disease index (OSDI) | Administered 4 weeks after
  The ocular surface disease index was assessed for ocular surface disease, including visual function (five items), eye symptoms (four items), and environmental factors (three items) , 0 point for no symptoms, 1 point for occasional symptoms, 2 points for symptoms of half a day, 3 points for most symptoms, and 4 points for symptoms during the whole day.
IOP(Intraocular pressure) | Administered 4, 12 weeks after
  IOP (fluid pressure inside the eye) was assessed using Goldmann applanation tonometry and measured in millimeters of mercury (mmHg). Data at 10:00 AM from Weeks 4, 8, and 12 were pooled. A more negative change indicates a greater amount of improvement. One eye (study eye) was subject to analysis.
Tear break up time (TBUT) | Administered 4, 12 weeks after
  After blinking blue fluorescein staining of the cobalt blue light source using a yellow filter, it was observed from the blinking point that there was a black spot, a streak pattern or a fluorine defect in the fluorescein-tear layer Was measured in seconds. The measurement results were repeated three times and average values were used.
Slit Lamp Biomicroscopy Findings - Limbal Redness | Administered 4, 12 weeks after
  Slit lamp Biomicroscopy findings will be assessed on Efron Grading scales scored to the nearest 0.1 on a scale of 0 - 4 (0=normal, 1=trace, 2=mild, 3=moderate, 4=severe).

CONTACTS AND LOCATIONS:
Locations (1):
- CHA University Bundang Medical Center, Seongnam, Bundang-gu, South Korea